CLINICAL TRIAL: NCT01102023
Title: Effect of Solar Salt Diet in Elderly Hypertensive Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Chung-Ang University Hosptial, Chung-Ang University College of Medicine (Other)
Collaborators: Mokpo National University (Other); the ministry of knowledge economy (Unknown)
Other Study IDs: C2009067(254)
Record Dates: First submitted 2010-04-08; First posted 2010-04-12 (Estimated); Last update posted 2010-04-12 (Estimated); Status verified 2010-03

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

ARMS (1):
- solar salt based-diet (Experimental)
  Interventions: Other: ordinary salt based- diet

INTERVENTIONS:
Other: ordinary salt based- diet

SUMMARY:
High sodium intake causes hypertension. Various efforts for reducing salt consumption are proceeding all over the world. Solar salt contains reduced sodium and abundant mineral, such as calcium, potassium, and magnesium, comparing to ordinary salt. Use of solar salt, instead of ordinary salt, may have beneficial effects to blood pressure.

The investigators are going to conduct a preliminary study that can support antihypertensive effect of solar salt intake.

ELIGIBILITY:
Inclusion Criteria:

* above 50 years elderly hypertensive patients
* possible oral intake

Exclusion Criteria:

* dementia, GDS>6
* terminal cancer patient

Min Age: 50 Years | Sex: All
Age Groups: Adult, Older Adult

PRIMARY OUTCOMES:
Blood pressure

CONTACTS AND LOCATIONS:
Locations (1):
- Lohas-clover silver hospital, Seoul, South Korea